CLINICAL TRIAL: NCT06192589
Title: Clinical Study to Evaluate Cannabidiol Liver Enzyme Elevations and Drug Interactions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SCR-016
Record Dates: First submitted 2023-12-18; First posted 2024-01-05 (Actual); Results first posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Cannabidiol; Drug Induced Liver Injury; Drug Interaction
Keywords: Cannabidiol; CBD; Liver enzyme elevation; Drug interactions
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — Cannabidiol; Citalopram; Morphine

STUDY DESIGN:
Intervention Model Description: This is a two-part study. Part 1 is a randomized, double-blind, placebo-controlled, parallel study in 200 subjects (150 subjects receiving cannabidiol and 50 subjects receiving placebo).
  Part 2 is an open-label, sequential study in 40 subjects (two separate cohorts of 20 subjects).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 of the study will be double-blind, and the blind will be maintained through a randomization schedule held by the dispensing pharmacist. The pharmacist (and designated staff member responsible for confirmation of study drug dose) will be unblinded to subject treatment assignment; however, the pharmacist will not perform any study procedures other than study drug preparation and dispensing.
  Part 2 is an open label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cannabidiol (Part 1) (Active Comparator): Subjects in this arm will receive oral solution cannabidiol at a dosage of 2.5 mg/kg twice a day, for a total of 5 mg/kg cannabidiol daily for 28 days.
  Interventions: Drug: Cannabidiol
- Placebo (Part 1) (Placebo Comparator): Subjects in this arm will receive oral solution placebo twice a day for 28 days.
  Interventions: Drug: Placebo
- Cannabidiol and Citalopram Drug Interaction (Part 2) (Active Comparator): Subjects in this arm will receive citalopram (20 mg) on Day 1 and Day 13 and oral solution cannabidiol at a dosage of 2.5 mg/kg twice a day (5 mg/kg cannabidiol daily) for 12 days (Day 6-17).
  Interventions: Drug: Cannabidiol; Drug: Citalopram
- Cannabidiol and Morphine Drug Interaction (Part 2) (Active Comparator): Subjects in this arm will receive morphine (15 mg) on Day 1, Day 4, and Day 11 and oral solution cannabidiol at a dosage of 2.5 mg/kg twice a day (5 mg/kg CBD daily) for 9 days (Day 4-12).
  Interventions: Drug: Cannabidiol; Drug: Morphine

INTERVENTIONS:
Drug: Cannabidiol — Cannabidiol (Epidiolex) will be administered orally 2.5 mg/kg twice daily (5 mg/kg/day) for 28 days in Part 1 and for 9 days (morphine cohort) or 12 days (citalopram cohort) in Part 2.
  Other Names: Epidiolex
  Arms: Cannabidiol (Part 1); Cannabidiol and Citalopram Drug Interaction (Part 2); Cannabidiol and Morphine Drug Interaction (Part 2)
Drug: Placebo — Placebo will be administered orally twice daily for 28 days in Part 1
  Arms: Placebo (Part 1)
Drug: Citalopram — Citalopram (Celexa) will be administered once at 20 mg on days 1 and 13.
  Other Names: Celexa
  Arms: Cannabidiol and Citalopram Drug Interaction (Part 2)
Drug: Morphine — Morphine will be administered once at 15 mg on days 1, 4, and 11.
  Arms: Cannabidiol and Morphine Drug Interaction (Part 2)

SUMMARY:
Cannabidiol (CBD) is available as a prescription drug product for the treatment of seizures associated with Lennox-Gastaut syndrome, Dravet syndrome, or tuberous sclerosis complex. At labeled doses up to 25 mg/kg/day, an increased risk of liver enzyme elevation and drug-induced liver injury has been observed. However, only limited evaluations of the risk of liver enzyme elevation of daily, lower dose CBD use are available. The potential for liver enzyme elevations with lower CBD doses with unapproved consumer products highlights a need for further research. In addition, CBD has the capacity to inhibit cytochrome P450 enzymes and uridine 5'-diphospho-glucuronosyltransferases, leading to potential drug-drug interactions with multiple common medications. The clinical significance of many of these interactions is also unclear. Furthermore, nonclinical studies have suggested the potential for CBD to cause reproductive and endocrine effects. As such, additional high-quality clinical pharmacology studies are needed to further characterize CBD's safety profile.

The objective of this study is to characterize the effects of daily CBD use at a dose within the range of what consumers are taking as unapproved CBD products on liver enzyme elevations, drug interactions, and endocrine measures.

DETAILED DESCRIPTION:
The cannabis plant contains bioactive compounds known as cannabinoids; delta-9 tetrahydrocannabinol (THC) and cannabidiol (CBD) are the most prevalent cannabinoids in most varieties of cannabis. The Agricultural Improvement Act (Farm Bill) of 2018 removed hemp, defined as cannabis and derivatives of cannabis with extremely low concentrations of THC, from the definition of marijuana in the Controlled Substances Act. Following this, many CBD products have been made available to consumers. However, hemp products remain subject to regulation under the Federal Food Drug & Cosmetic Act, when applicable (e.g., as drugs, foods, dietary supplements, cosmetics, veterinary products) and the growing CBD products market raises various safety concerns, especially with long-term use.

CBD is available as a prescription drug product for the treatment of seizures associated with Lennox-Gastaut syndrome, Dravet syndrome, or tuberous sclerosis complex. At labeled doses up to 25 mg/kg/day, an increased risk of liver enzyme elevation and drug-induced liver injury has been observed. However, only limited evaluations of the risk of liver enzyme elevation of daily, lower dose CBD use are available. The potential for liver enzyme elevations with CBD doses in unapproved consumer products highlights a need for further research to quantify risks at these doses. In addition, CBD has the capacity to inhibit cytochrome P450 enzymes and uridine 5'-diphospho-glucuronosyltransferases, leading to potential drug-drug interactions with multiple common medications. The clinical significance of many of these interactions is also unclear. Furthermore, nonclinical studies have suggested the potential for CBD to cause reproductive and endocrine effects. As such, additional high-quality clinical pharmacology studies are needed to further characterize CBD's safety profile.

This study will be divided into two parts.

In Part 1, 200 healthy subjects will be randomized to 5 mg/kg/day of CBD (150 subjects) or placebo (50 subjects) for 4 weeks with weekly laboratory assessments to characterize the percentage of participants with liver enzyme elevation (primary endpoint) or meeting withdrawal criteria for potential drug-induced liver injury (secondary endpoint). Additional secondary endpoints include the change from baseline after 4 weeks of daily CBD dosing for male reproductive (testosterone and inhibin B) and thyroid hormones (thyroid stimulating hormone [TSH], triiodothyronine [T3] and thyroxine [T4]) as secondary endpoints. Exploratory endpoints include additional characterization of liver findings and other blood biomarkers.

In Part 2, 40 healthy subjects will receive either oral citalopram (20 subjects) or morphine (20 subjects) at baseline and then again after receiving CBD 5 mg/kg/day to characterize the effect of daily cannabidiol use on the plasma concentration of citalopram and morphine. Citalopram was selected because it is a common prescription medication for depression and anxiety that is metabolized by CYP2C19 and CYP3A4, which CBD inhibits. Morphine was selected because it is a common opioid analgesic that is metabolized by UGT2B7, which CBD inhibits.

ELIGIBILITY:
Inclusion Criteria:

1. Subject signs an institutional review board (IRB) approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act authorization) before any study related procedures are performed.
2. Subject is a healthy, non-smoking man or woman, 18 to 55 years of age, inclusive, who weighs at least 50 kg (110 lbs) and has a body mass index of 18.5 to 33.0 kg/m2, inclusive, at Screening and check-in (Day -1).
3. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, 12-lead ECG results, and physical examination findings at screening or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee).
4. Subject must have a negative test result for alcohol and illicit drugs at screening and check-in (Day -1).
5. Participants must agree to refrain from using any of the following for the duration of the study: alcohol, nicotine containing products, marijuana or marijuana-derived products, hemp or hemp-derived products, including CBD (except for provided study drug), and illicit drugs of any kind.
6. Subject must test negative for severe acute respiratory syndrome corona virus 2 (SARS-CoV-2) by a rapid antigen test at check-in for all study periods. If a subject's test comes back as invalid, the test can be repeated.
7. Female subjects must be of non-childbearing potential (non-childbearing potential includes post-menopausal females defined as spontaneous amenorrhea for at least 12 months with FSH in the post-menopausal range and females who have undergone a hysterectomy) or, if they are of childbearing potential, they must: 1) have negative serum HCG at screening and check-in 2) have been strictly abstinent for 1 month before check-in (Day -1) and agree to remain strictly abstinent for the duration of the study and for at least 1 month after the last application of study drug; OR 3) be practicing 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from Screening until at least 1 month after the end of the study.
8. Male subjects must agree to practice 2 highly effective methods of birth control (as determined by the investigator or designee) beginning at check-in (Day -1) until at least 3 months after the last dose of study drug. Male subjects may not donate sperm for 90 days after the end of the study.
9. Subject agrees to and is highly likely (as determined by the investigator) to comply with the protocol defined procedures and to complete the study.

Exclusion Criteria:

1. Abnormal liver labs at screening on check-in (Day -1), defined as any of the following (tests may be repeated once for confirmation at screening and check-in):

   1. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 × ULN. (The ULN for ALT will be 33 U/L for males and 25 U/L for females.)
   2. Total bilirubin (TBL) > ULN.
   3. International normalized ratio (INR) > 1.3
2. Use or intend to use any medications/products in the 14 days prior to check-in (Day -1), unless deemed acceptable by the investigator
3. Subject is currently participating in another clinical study of an investigational drug or has been treated with any investigational drug within 30 days or 5 half-lives (whichever is longer) of dosing for this study.
4. Subject has used nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, electronic cigarettes) within 6 weeks of Screening. Subjects must refrain from using these throughout the study.
5. Subject has consumed alcohol, xanthine-containing products (e.g., tea, coffee, chocolate, cola), caffeine, kava melatonin, St Johns Wart, grapefruit, or grapefruit juice within 24 hours of check-in. Subjects must refrain from ingesting these throughout the study.
6. Subject is unable to tolerate a controlled, quiet study conduct environment, including avoidance of music, television, movies, games, and activities that may cause excitement, emotional tension, or arousal during the prespecified time points (e.g., before and during CBD dosing).
7. Subject has a history of consuming more than 14 units of alcoholic beverages per week within 6 months before Screening, has a history of alcoholism or drug/chemical/substance abuse within 2 years before Screening (Note: 1 unit = 12 ounces of beer, 4 ounces of wine, or 1 ounce of spirits/hard liquor)
8. Subject has a positive test result for alcohol or drugs of misuse (amphetamines, barbiturates, benzodiazepines, cocaine, alcohol, opiates, phencyclidine, propoxyphene, and methadone) at Screening or Check-in (Day -1 [both Parts]; Day 10 [Part 2, morphine DDI]; Day 12 [Part 2, citalopram DDI]).
9. Subject has a positive test result for cannabinoids (THC) at screening or Day -1.
10. Subject has a history of opioid or narcotic misuse.
11. Subject has a history of suicidal ideation or previous suicide attempts
12. Subject has a history or evidence of a clinically significant disorder, condition, or disease (e.g., cancer, human immunodeficiency virus [HIV], hepatic or renal impairment) that, in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
13. Subject has any signs or symptoms that are consistent with Coronavirus Disease 2019 (COVID-19) per Center for Disease Control (CDC) recommendations at screening or check-in (Day -1). These include subjects with fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, or diarrhea may have COVID-19. In addition, the subject has any other findings suggestive of COVID-19 risk in the opinion of the investigator.
14. Subject has known or suspected allergies or sensitivities to the study drug or placebo components (e.g., sucralose, sesame).
15. Subjects with a documented hypersensitivity reaction to cannabidiol
16. Subjects with a documented medical history of clinical disorders related to mood, anxiety or panic, including diagnosed depression, generalized anxiety disorder or panic attacks.
17. Subject has any condition possibly affecting study drug absorption (e.g., gastrectomy, Crohn's disease, irritable bowel syndrome). Uncomplicated cholecystectomies and appendectomies may be included at the investigator's discretion.
18. Subject has clinical laboratory test results (hematology, serum chemistry and urinalysis) at Screening or Check-In that are outside the reference ranges provided by the clinical laboratory and considered clinically significant by the investigator. Tests may be repeated once for confirmation at both Screening and Check-In.
19. Subject has a positive test result at Screening for HIV 1 or 2 antibody, hepatitis C virus antibodies, or hepatitis B surface antigen.
20. Subject has a mean systolic blood pressure <85 or >145 mmHg or a mean diastolic blood pressure <45 or >95 mmHg at either Screening or Check-in. Blood pressure will be measured in triplicate after the subject has been resting in a supine position for a minimum of 5 minutes.
21. Subject is unable or unwilling to undergo multiple venipunctures for blood sample collection because of poor tolerability or is unlikely to complete the study due to poor venous access.
22. Female subject is currently pregnant or lactating or was within 3 months of the study.
23. Subject has had any significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days, or donated plasma within 7 days before Check-in.
24. Subject has any other condition that precludes his or her participation in the study (as determined by the investigator).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 241 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Fein, MD, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan is to make data from the study publicly available as part of a manuscript publication. In addition, the protocol and statistical analysis plan will be made available online at this site as well as with any eventual publications.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available at the time of manuscript publication.
Access Criteria: No restrictions.

REFERENCES:
- [Background] 1. U.S. Food and Drug Administration (FDA) Science Board. (2022, June 3). Background materials for the June 14, 2022 meeting of the Science Board to the FDA. Retrieved from https://www.fda.gov/advisory-committees/advisory-committee-roster/science-board-fda/2022-meetings#event-materials.
- [Background] 2. Cannabidiol (Epidiolex ®) oral solution label obtained from https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/210365lbl.pdf
- [Background] Lo LA, Christiansen A, Eadie L, Strickland JC, Kim DD, Boivin M, Barr AM, MacCallum CA. Cannabidiol-associated hepatotoxicity: A systematic review and meta-analysis. J Intern Med. 2023 Jun;293(6):724-752. doi: 10.1111/joim.13627. Epub 2023 Mar 13. PMID 36912195
- [Background] Crippa JAS, Zuardi AW, Guimaraes FS, Campos AC, de Lima Osorio F, Loureiro SR, Dos Santos RG, Souza JDS, Ushirohira JM, Pacheco JC, Ferreira RR, Mancini Costa KC, Scomparin DS, Scarante FF, Pires-Dos-Santos I, Mechoulam R, Kapczinski F, Fonseca BAL, Esposito DLA, Pereira-Lima K, Sen S, Andraus MH, Hallak JEC; Burnout and Distress Prevention With Cannabidiol in Front-line Health Care Workers Dealing With COVID-19 (BONSAI) Trial Investigators. Efficacy and Safety of Cannabidiol Plus Standard Care vs Standard Care Alone for the Treatment of Emotional Exhaustion and Burnout Among Frontline Health Care Workers During the COVID-19 Pandemic: A Randomized Clinical Trial. JAMA Netw Open. 2021 Aug 2;4(8):e2120603. doi: 10.1001/jamanetworkopen.2021.20603. PMID 34387679
- [Background] 5. U.S. Food and Drug Administration (FDA). Clinical Pharmacology and Biopharmaceutics Review. Retrieved from https://www.accessdata.fda.gov/drugsatfda_docs/nda/2018/210365Orig1s000ClinPharmR.pdf
- [Background] 6. EFSA NDA Panel (EFSA Panel on Nutrition, Novel Foods and Food Allergens), Turck, D, Bohn, T, Castenmiller, J, De Henauw, S, Hirsch-Ernst, KI, Maciuk, A, Mangelsdorf, I, McArdle, HJ, Naska, A, Pelaez, C, Pentieva, K, Siani, A, Thies, F, Tsabouri, S, Vinceti, M, Cubadda, F, Frenzel, T, Heinonen, M, Marchelli, R, Neuhäuser-Berthold, M, Poulsen, M, Prieto Maradona, M, Schlatter, JR, Trezza, V, van Loveren, H, Albert, O, Dumas, C, Germini, A, Gelbmann, W, Kass, G, Kouloura, E, Noriega Fernandez, E, Rossi, A and Knutsen, HK, 2022. Statement on safety of cannabidiol as a novel food: data gaps and uncertainties. EFSA Journal 2022; 20(6):7322, 25 pp. https://doi.org/10.2903/j.efsa.2022.7322
- [Background] Carvalho RK, Andersen ML, Mazaro-Costa R. The effects of cannabidiol on male reproductive system: A literature review. J Appl Toxicol. 2020 Jan;40(1):132-150. doi: 10.1002/jat.3831. Epub 2019 Jul 17. PMID 31313338
- [Background] Tallon MJ, Child R. Subchronic oral toxicity assessment of a cannabis extract. Regul Toxicol Pharmacol. 2023 Oct;144:105496. doi: 10.1016/j.yrtph.2023.105496. Epub 2023 Sep 19. PMID 37734651
- [Background] Anderson LL, Doohan PT, Oldfield L, Kevin RC, Arnold JC, Berger M, Amminger GP, McGregor IS. Citalopram and Cannabidiol: In Vitro and In Vivo Evidence of Pharmacokinetic Interactions Relevant to the Treatment of Anxiety Disorders in Young People. J Clin Psychopharmacol. 2021 Sep-Oct 01;41(5):525-533. doi: 10.1097/JCP.0000000000001427. PMID 34121064
- [Background] Armstrong SC, Cozza KL. Pharmacokinetic drug interactions of morphine, codeine, and their derivatives: theory and clinical reality, part I. Psychosomatics. 2003 Mar-Apr;44(2):167-71. doi: 10.1176/appi.psy.44.2.167. PMID 12618536
- [Background] 11. Citalopram (Celexa ®) tablet label obtained from https://www.accessdata.fda.gov/drugsatfda_docs/label/2022/020822s041lbl.pdf
- [Background] 12. Morphine Sulfate tablet label obtained from https://www.accessdata.fda.gov/drugsatfda_docs/label/2021/022207s010lbl.pdf
- [Background] Iannone LF, Arena G, Battaglia D, Bisulli F, Bonanni P, Boni A, Canevini MP, Cantalupo G, Cesaroni E, Contin M, Coppola A, Cordelli DM, Cricchiuti G, De Giorgis V, De Leva MF, De Rinaldis M, d'Orsi G, Elia M, Galimberti CA, Morano A, Granata T, Guerrini R, Lodi MAM, La Neve A, Marchese F, Masnada S, Michelucci R, Nosadini M, Pilolli N, Pruna D, Ragona F, Rosati A, Santucci M, Spalice A, Pietrafusa N, Striano P, Tartara E, Tassi L, Papa A, Zucca C, Russo E, Mecarelli O; CBD LICE Italy Study Group. Results From an Italian Expanded Access Program on Cannabidiol Treatment in Highly Refractory Dravet Syndrome and Lennox-Gastaut Syndrome. Front Neurol. 2021 May 20;12:673135. doi: 10.3389/fneur.2021.673135. eCollection 2021. PMID 34093420
- [Background] Sharbaf Shoar N, Fariba KA, Padhy RK. Citalopram. 2023 Nov 7. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482222/ PMID 29489221
- [Background] Aithal GP, Watkins PB, Andrade RJ, Larrey D, Molokhia M, Takikawa H, Hunt CM, Wilke RA, Avigan M, Kaplowitz N, Bjornsson E, Daly AK. Case definition and phenotype standardization in drug-induced liver injury. Clin Pharmacol Ther. 2011 Jun;89(6):806-15. doi: 10.1038/clpt.2011.58. Epub 2011 May 4. PMID 21544079
- [Background] Arnold JC, McCartney D, Suraev A, McGregor IS. The safety and efficacy of low oral doses of cannabidiol: An evaluation of the evidence. Clin Transl Sci. 2023 Jan;16(1):10-30. doi: 10.1111/cts.13425. Epub 2022 Oct 19. PMID 36259271
- [Derived] Florian J, Salcedo P, Burkhart K, Shah A, Chekka LMS, Keshishi D, Patel V, Yang S, Fein M, DePalma R, Matta M, Strauss DG, Rouse R. Cannabidiol and Liver Enzyme Level Elevations in Healthy Adults: A Randomized Clinical Trial. JAMA Intern Med. 2025 Sep 1;185(9):1070-1078. doi: 10.1001/jamainternmed.2025.2366. PMID 40622698

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cannabidiol (Part 1) | Placebo (Part 1) | Cannabidiol and Citalopram Drug Interaction (Part 2) | Cannabidiol and Morphine Drug Interaction (Part 2)
Started | 151 | 50 | 20 | 20
Completed | 133 | 47 | 20 | 18
Not Completed | 18 | 3 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Citalopram and Cannabidiol (Part 2): Subjects in this arm will receive citalopram (20 mg) on Day 1 and Day 13 and oral solution cannabidiol at a dosage of 2.5 mg/kg twice a day (5 mg/kg cannabidiol daily) for 12 days (Day 6-17).
  Cannabidiol: Cannabidiol (Epidiolex) will be administered orally 2.5 mg/kg twice daily (5 mg/kg/day) for 28 days in Part 1 and for 9 days (morphine cohort) or 12 days (citalopram cohort) in Part 2.
  Citalopram: Citalopram (Celexa) will be administered once at 20 mg on days 1 and 13.
- Morphine and Cannabidiol (Part 2): Subjects in this arm will receive morphine (15 mg) on Day 1 (baseline), Day 4, and Day 11 (with CBD). Oral solution cannabidiol at a dosage of 2.5 mg/kg twice a day (5 mg/kg cannabidiol daily) for 9 days (Day 4-12).
  Cannabidiol: Cannabidiol (Epidiolex) will be administered orally 2.5 mg/kg twice daily (5 mg/kg/day) for 28 days in Part 1 and for 9 days (morphine cohort) or 12 days (citalopram cohort) in Part 2.
  Morphine: Morphine sulfate tablet will be administered once at 15 mg on days 1, 4 and 11.
- Total: Total of all reporting groups
Arm/Group | Cannabidiol (Part 1) | Placebo (Part 1) | Citalopram and Cannabidiol (Part 2) | Morphine and Cannabidiol (Part 2) | Total
Number analyzed (Participants) | 151 | 50 | 20 | 20 | 241
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [31 to 44] | 32 [29 to 41] | 37 [29 to 49] | 38 [35 to 44] | 36 [30.5 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 21 | 7 | 8 | 104
  Male | 83 | 29 | 13 | 12 | 137
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 3 | 3 | 0 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 64 | 23 | 9 | 8 | 104
  White | 77 | 22 | 8 | 10 | 117
  More than one race | 2 | 1 | 1 | 1 | 5
  Unknown or Not Reported | 4 | 1 | 2 | 0 | 7
Median Body Weight [Median (Full Range); unit: kg] | 80.2 [50.6 to 110.0] | 75.9 [53.0 to 103.0] | 79.5 [59.6 to 102.1] | 82.7 [58.9 to 102] | 80.1 [50.6 to 110.0]
Median Height [Median (Full Range); unit: m] | 1.71 [1.53 to 1.94] | 1.72 [1.52 to 1.87] | 1.74 [1.54 to 1.87] | 1.76 [1.53 to 1.90] | 1.72 [1.52 to 1.94]
Median Body Mass Index [Median (Full Range); unit: kg/m2] | 27.1 [18.6 to 33] | 26 [19.2 to 32] | 26.6 [21.7 to 32.1] | 26.7 [22.1 to 32.3] | 26.7 [18.6 to 33]

OUTCOME MEASURES:

1. Primary Outcome: Part 1 - Percentage of Participants With an Alanine Transaminase (ALT) or Aspartate Aminotransferase (AST) Liver Enzyme Elevation Greater Than Three Times the Upper Limit of Normal (> 3 × ULN).
Description: The upper limit of normal (ULN), based on consensus criteria, for the liver transaminase ALT (Alanine transaminase) is defined as 33 U/L for males and 25 U/L for females. An ALT evaluation three times the ULN for males would be 99 U/L and 75 U/L for females.
Time Frame: Days 1 through 35
Population: The liver safety analysis population will include all subjects who receive at least 1 dose of the study drug and have at least one on-treatment liver and hematology lab assessment. Subjects in the liver safety analysis population will be used for the planned primary, secondary, and exploratory analyses related to liver enzyme elevations and liver events. Results will be reported as percentages with a 95% confidence interval (CI) based on a Kaplan-Meier analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cannabidiol (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 151 | 50
percentage of participants | 5.6 [1.8 to 9.3] | 0 [0 to 7.6]

2. Primary Outcome: Part 2 - Area Under the Plasma Concentration-time Curve (AUC) of Citalopram When Administered Alone Versus When Co-administered With Cannabidiol After 7 Days of CBD Dosing.
Description: AUC will be determined by collecting pharmacokinetic (PK) blood samples and calculated using noncompartmental analysis. 13 PK samples will be obtained with each citalopram dose for a total number of 26 PK samples per citalopram cohort participant. The outcome measure reported will be the geometric mean ratio for citalopram alone compared to citalopram after 7 days of CBD dosing.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hours after each citalopram dose (Days 1 and 13)
Population: All subjects who receive at least one dose of study drug and have at least one on-treatment PK sample collected. One subject was removed from the analysis due to a protocol violation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Part 2: Citalopram: Subjects in this arm will receive citalopram (20 mg) on Day 1 and Day 13 and oral solution cannabidiol at a dosage of 2.5 mg/kg twice a day (5 mg/kg cannabidiol daily) for 12 days (Day 6-17).
  Reported data is for citalopram exposures from citalopram alone (Day 1-5).
- Part 2: Citalopram and Cannabidiol: Subjects in this arm will receive citalopram (20 mg) on Day 1 and Day 13 and oral solution cannabidiol at a dosage of 2.5 mg/kg twice a day (5 mg/kg cannabidiol daily) for 12 days (Day 6-17).
  Reported data is for citalopram exposures from citalopram (Day 13-17) coadministered with cannabidiol.
Arm/Group | Part 2: Citalopram | Part 2: Citalopram and Cannabidiol
Number analyzed (Participants) | 19 | 19
ng*hr/mL | 1033 (26) | 1475 (24)
Statistical Analysis 1: Comparison: Part 2: Citalopram vs Part 2: Citalopram and Cannabidiol; Area under the curve was log-transformed and the values between groups were compared using a linear mixed effects model with group as a categorical variable and subject as a random effect; Test type: Other — A difference in exposure was concluded if the 2-sided 90% CI of the geometric mean ratio excluded 1, which is standard in pharmacokinetic studies; p < 0.01, Mixed Models Analysis — Analyses are not adjusted for multiplicity; Geometric mean ratio = 1.43, 90% CI 2-sided [1.34 to 1.52] — Comparison was the effect of cannabidiol on citalopram compared to citalopram alone

3. Primary Outcome: Part 2 - Maximum Concentration (Cmax) of Citalopram When Administered Alone Versus When Co-administered With CBD After 7 Days of Cannabidiol Dosing.
Description: Cmax will be determined by collecting pharmacokinetic (PK) blood samples and calculated using noncompartmental analysis. 13 PK samples will be obtained with each citalopram dose for a total number of 26 PK samples per citalopram cohort participant. The outcome measure reported will be the geometric mean ratio for citalopram alone compared to citalopram after 7 days of CBD dosing.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hours after each citalopram dose (Days 1 and 13)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: Citalopram | Part 2: Citalopram and Cannabidiol
Number analyzed (Participants) | 19 | 19
ng/mL | 23 (21) | 26 (24)
Statistical Analysis 1: Comparison: Part 2: Citalopram vs Part 2: Citalopram and Cannabidiol; Maximum concentration was log-transformed and the values between groups were compared using a linear mixed effects model with group as a categorical variable and subject as a random effect; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.01, Mixed Models Analysis — Analyses are not adjusted for multiplicity; Geometric mean ratio = 1.12, 90% CI 2-sided [1.06 to 1.17] — Comparison was the effect of cannabidiol on citalopram compared to citalopram alone

4. Primary Outcome: Part 2 - Morphine AUC When Administered Alone Versus When Co-administered With the First Dose of Cannabidiol and After 7 Days of CBD Dosing.
Description: AUC will be determined by collecting pharmacokinetic (PK) blood samples and calculated using noncompartmental analysis.13 PK samples will be obtained with each morphine dose for a total number of 39 PK samples per morphine cohort participant. The outcome measure reported will be the geometric mean ratio for morphine alone compared to morphine after 7 days of CBD dosing.
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 12, 24, and 48 hours after each morphine dose (Days 1, 4, and 11)
Population: All subjects who receive at least one dose of study drug and have at least one on-treatment PK sample collected. For morphine and its metabolites, number of subjects is 20 for morphine alone and morphine with a single dose of CBD. For morphine with multiple doses of CBD, the sample size is 18 as two subjects discontinued from the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Part 2: Morphine: Subjects in this arm will receive morphine (15 mg) on Day 1 (baseline), Day 4, and Day 11 (with CBD). Oral solution cannabidiol at a dosage of 2.5 mg/kg twice a day (5 mg/kg cannabidiol daily) for 9 days (Day 4-12).
  Reported data is for morphine exposures from morphine alone (Day 1-2).
- Part 2: Morphine and Single Dose Cannabidiol: Subjects in this arm will receive morphine (15 mg) on Day 1 (baseline), Day 4, and Day 11 (with CBD). Oral solution cannabidiol at a dosage of 2.5 mg/kg twice a day (5 mg/kg cannabidiol daily) for 9 days (Day 4-12).
  Reported data is for morphine exposures from morphine with a single dose of cannabidiol (Day 4-5).
- Part 2: Morphine and Multiple Doses of Cannabidiol: Subjects in this arm will receive morphine (15 mg) on Day 1 (baseline), Day 4, and Day 11 (with CBD). Oral solution cannabidiol at a dosage of 2.5 mg/kg twice a day (5 mg/kg cannabidiol daily) for 9 days (Day 4-12).
  Reported data is for morphine exposures from morphine following multiple doses of cannabidiol (Day 11-12).
Arm/Group | Part 2: Morphine | Part 2: Morphine and Single Dose Cannabidiol | Part 2: Morphine and Multiple Doses of Cannabidiol
Number analyzed (Participants) | 20 | 20 | 18
ng*hr/mL | 44 (45) | 47 (51) | 51 (60)
Statistical Analysis 1: Comparison: Part 2: Morphine vs Part 2: Morphine and Single Dose Cannabidiol; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.34, Mixed Models Analysis; Analyses are not adjusted for multiplicity; Geometric mean ratio = 1.06, 90% CI 2-sided [0.96 to 1.16] — Comparison was the effect of a single dose of cannabidiol on morphine compared to morphine alone
Statistical Analysis 2: Comparison: Part 2: Morphine vs Part 2: Morphine and Multiple Doses of Cannabidiol; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.10, Mixed Models Analysis; Analyses are not adjusted for multiplicity; Geometric mean ratio = 1.12, 90% CI 2-sided [1.00 to 1.26] — Comparison was the effect of a multiple doses of cannabidiol on morphine compared to morphine alone

5. Primary Outcome: Part 2 - Morphine Cmax When Administered Alone Versus When Co-administered With the First Dose of Cannabidiol and After 7 Days of Cannabidiol Dosing.
Description: Cmax will be determined by collecting pharmacokinetic (PK) blood samples and calculated using noncompartmental analysis.13 PK samples will be obtained with each morphine dose for a total number of 39 PK samples per morphine cohort participant. The outcome measure reported will be the geometric mean ratio for morphine alone compared to morphine after 7 days of CBD dosing.
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 12, 24, and 48 hours after each morphine dose (Days 1, 4, and 11)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: Morphine | Part 2: Morphine and Single Dose Cannabidiol | Part 2: Morphine and Multiple Doses of Cannabidiol
Number analyzed (Participants) | 20 | 20 | 18
ng/mL | 8.3 (40) | 9.9 (45) | 9.3 (31)
Statistical Analysis 1: Comparison: Part 2: Morphine vs Part 2: Morphine and Single Dose Cannabidiol; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.02, Mixed Models Analysis; Analyses are not adjusted for multiplicity; Geometric mean ratio = 1.19, 90% CI 2-sided [1.05 to 1.35] — Comparison was the effect of a single dose of cannabidiol on morphine compared to morphine alone
Statistical Analysis 2: Comparison: Part 2: Morphine vs Part 2: Morphine and Multiple Doses of Cannabidiol; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.29, Mixed Models Analysis; Analyses are not adjusted for multiplicity; Geometric mean ratio = 1.11, 90% CI 2-sided [0.94 to 1.30] — Comparison was the effect of multiple doses of cannabidiol on morphine compared to morphine alone

6. Secondary Outcome: Part 1 - Percentage of Participants Meeting Withdrawal Criteria for Potential Drug-induced Liver Injury (DILI).
Description: Withdrawal criteria for potential drug-induced liver-injury: laboratory results meeting any of the following criteria.
  * ALT or AST > 3 x ULN (ULN for ALT is 33 U/L for males and 25 U/L for females) with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%) OR
  * ALT elevation ≥ 5 × ULN (ULN for ALT is 33 U/L for males and 25 U/L for females) OR
  * Alkaline phosphatase (ALP) elevation ≥ 2 × ULN (with accompanying elevations of gamma-glutamyl transpeptidase (GGT) in the absence of known bone pathology driving the rise in ALP level) OR
  * ALT elevation ≥ 3 × ULN and bilirubin concentration > 2 × ULN
Time Frame: Days 1 through 35
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cannabidiol (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 151 | 50
percentage of participants | 4.9 [1.3 to 8.4] | 0 [0 to 7.6]

7. Secondary Outcome: Part 1 - Change From Baseline in Total Testosterone in Male Participants After Cannabidiol Administration Compared to Placebo.
Description: Endocrine assessments for total testosterone will be obtained through blood samples. A linear mixed effect model will be utilized to obtain least squares means for each treatment group.
Time Frame: Days 1 and 29
Population: Analyses include male participants with time-matched samples at day 1 and 29
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/dL
Arm/Group | Cannabidiol (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 26
ng/dL | 5.0 [-20.0 to 30.0] | -13.6 [-57.1 to 29.9]

8. Secondary Outcome: Part 1 - Change From Baseline in Inhibin B in Male Participants After Cannabidiol Administration Compared to Placebo.
Description: Endocrine assessments for inhibin B will be obtained through blood samples. A linear mixed effect model will be utilized to obtain least squares means for each treatment group.
Time Frame: Days 1 and 29
Population: Analyses include male participants with time-matched samples at day 1 and 29
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Cannabidiol (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 77 | 26
pg/mL | 5.8 [0.8 to 10.7] | 8.2 [-0.0 to 16.5]

9. Secondary Outcome: Part 1 - Change From Baseline in Thyroid Stimulating Hormone (TSH) After Cannabidiol Administration Compared to Placebo.
Description: Endocrine assessments for TSH will be obtained through blood samples. A linear mixed effect model will be utilized to obtain least squares means for each treatment group.
Time Frame: Days 1 and 29
Population: Analyses include all participants with time-matched samples at day 1 and 29. Participants without day 29 samples (e.g., discontinued treatment prior to day 29) were excluded from the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: mU/mL
Arm/Group | Cannabidiol (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 139 | 47
mU/mL | 0.073 [-0.003 to 0.148] | 0.005 [-0.124 to 0.134]

10. Secondary Outcome: Part 1 - Change From Baseline in Total T3 After Cannabidiol Administration Compared to Placebo.
Description: Endocrine assessments for total T3 will be obtained through blood samples. A linear mixed effect model will be utilized to obtain least squares means for each treatment group.
Time Frame: Days 1 and 29
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cannabidiol (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 139 | 47
ng/mL | -0.006 [-0.023 to 0.011] | 0.014 [-0.015 to 0.043]

11. Secondary Outcome: Part 1 - Change From Baseline in Free T4 After Cannabidiol Administration Compared to Placebo.
Description: Endocrine assessments for free T4 will be obtained through blood samples. A linear mixed effect model will be utilized to obtain least squares means for each treatment group.
Time Frame: Days 1 and 29
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cannabidiol (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 139 | 47
ng/mL | -0.014 [-0.025 to -0.003] | -0.012 [-0.031 to 0.006]

12. Secondary Outcome: Part 2 - Morphine-3-glucuronide (M3G) AUC When Morphine is Administered Alone Versus When Co-administered With Cannabidiol.
Description: AUC will be determined by collecting pharmacokinetic (PK) blood samples and calculated using noncompartmental analysis.13 PK samples will be obtained with each morphine dose for a total number of 39 PK samples per morphine cohort participant. The outcome measure reported will be the geometric mean ratio for morphine-3-glucuronide (M3G) alone compared to morphine-3-glucuronide (M3G) after 7 days of CBD dosing.
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 12, 24, and 48 hours after each morphine dose (Days 1, 4, and 11)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Part 2: Morphine: Subjects in this arm will receive morphine (15 mg) on Day 1 (baseline), Day 4, and Day 11 (with CBD). Oral solution cannabidiol at a dosage of 2.5 mg/kg twice a day (5 mg/kg cannabidiol daily) for 9 days (Day 4-12).
  Reported data is for M3G exposures from morphine alone (Day 1-2).
- Part 2: Morphine and Single Dose Cannabidiol: Subjects in this arm will receive morphine (15 mg) on Day 1 (baseline), Day 4, and Day 11 (with CBD). Oral solution cannabidiol at a dosage of 2.5 mg/kg twice a day (5 mg/kg cannabidiol daily) for 9 days (Day 4-12).
  Reported data is for M3G exposures from morphine with a single dose of cannabidiol (Day 4-5).
- Part 2: Morphine and Multiple Doses of Cannabidiol: Subjects in this arm will receive morphine (15 mg) on Day 1 (baseline), Day 4, and Day 11 (with CBD). Oral solution cannabidiol at a dosage of 2.5 mg/kg twice a day (5 mg/kg cannabidiol daily) for 9 days (Day 4-12).
  Reported data is for M3G exposures from morphine following multiple doses of cannabidiol (Day 11-12).
Arm/Group | Part 2: Morphine | Part 2: Morphine and Single Dose Cannabidiol | Part 2: Morphine and Multiple Doses of Cannabidiol
Number analyzed (Participants) | 20 | 20 | 18
ng*hr/mL | 2416 (18) | 2450 (17) | 2382 (14)
Statistical Analysis 1: Comparison: Part 2: Morphine vs Part 2: Morphine and Single Dose Cannabidiol; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.47, Mixed Models Analysis; Analyses are not adjusted for multiplicity; Geometric mean ratio = 1.01, 90% CI 2-sided [0.98 to 1.05] — Comparison was the effect of a single dose of cannabidiol on morphine compared to morphine alone
Statistical Analysis 2: Comparison: Part 2: Morphine vs Part 2: Morphine and Multiple Doses of Cannabidiol; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.73, Mixed Models Analysis; Analyses are not adjusted for multiplicity; Geometric mean ratio = 0.99, 90% CI 2-sided [0.96 to 1.03] — Comparison was the effect of multiple doses of cannabidiol on morphine compared to morphine alone

13. Secondary Outcome: Part 2 - M3G Cmax When Morphine is Administered Alone Versus When Co-administered With Cannabidiol.
Description: Cmax will be determined by collecting pharmacokinetic (PK) blood samples and calculated using noncompartmental analysis.13 PK samples will be obtained with each morphine dose for a total number of 39 PK samples per morphine cohort participant. The outcome measure reported will be the geometric mean ratio for morphine-3-glucuronide (M3G) alone compared to morphine-3-glucuronide (M3G) after 7 days of CBD dosing.
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 12, 24, and 48 hours after each morphine dose (Days 1, 4, and 11)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: Morphine | Part 2: Morphine and Single Dose Cannabidiol | Part 2: Morphine and Multiple Doses of Cannabidiol
Number analyzed (Participants) | 20 | 20 | 18
ng/mL | 265 (21) | 296 (29) | 256 (25)
Statistical Analysis 1: Comparison: Part 2: Morphine vs Part 2: Morphine and Single Dose Cannabidiol; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.03, Mixed Models Analysis; Analyses are not adjusted for multiplicity; Geometric mean ratio = 1.12, 90% CI 2-sided [1.03 to 1.21] — Comparison was the effect of a single dose of cannabidiol on morphine compared to morphine alone
Statistical Analysis 2: Comparison: Part 2: Morphine vs Part 2: Morphine and Multiple Doses of Cannabidiol; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.66, Mixed Models Analysis; Analyses are not adjusted for multiplicity; Geometric mean ratio = 0.98, 90% CI 2-sided [0.91 to 1.06] — Comparison was the effect of multiple doses of cannabidiol on morphine compared to morphine alone

14. Secondary Outcome: Part 2 - Morphine-6-glucuronide (M6G) AUC When Morphine is Administered Alone Versus When Co-administered With Cannabidiol.
Description: AUC will be determined by collecting pharmacokinetic (PK) blood samples and calculated using noncompartmental analysis.13 PK samples will be obtained with each morphine dose for a total number of 39 PK samples per morphine cohort participant. The outcome measure reported will be the geometric mean ratio for morphine-6-glucuronide (M6G) alone compared to morphine-6-glucuronide (M6G) after 7 days of CBD dosing.
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 12, 24, and 48 hours after each morphine dose (Days 1, 4, and 11)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Part 2: Morphine: Subjects in this arm will receive morphine (15 mg) on Day 1 (baseline), Day 4, and Day 11 (with CBD). Oral solution cannabidiol at a dosage of 2.5 mg/kg twice a day (5 mg/kg cannabidiol daily) for 9 days (Day 4-12).
  Reported data is for M6G exposures from morphine alone (Day 1-2).
- Part 2: Morphine and Single Dose Cannabidiol: Subjects in this arm will receive morphine (15 mg) on Day 1 (baseline), Day 4, and Day 11 (with CBD). Oral solution cannabidiol at a dosage of 2.5 mg/kg twice a day (5 mg/kg cannabidiol daily) for 9 days (Day 4-12).
  Reported data is for M6G exposures from morphine with a single dose of cannabidiol (Day 4-5).
- Part 2: Morphine and Multiple Doses of Cannabidiol: Subjects in this arm will receive morphine (15 mg) on Day 1 (baseline), Day 4, and Day 11 (with CBD). Oral solution cannabidiol at a dosage of 2.5 mg/kg twice a day (5 mg/kg cannabidiol daily) for 9 days (Day 4-12).
  Reported data is for M6G exposures from morphine following multiple doses of cannabidiol (Day 11-12).
Arm/Group | Part 2: Morphine | Part 2: Morphine and Single Dose Cannabidiol | Part 2: Morphine and Multiple Doses of Cannabidiol
Number analyzed (Participants) | 20 | 20 | 18
ng*hr/mL | 327 (30) | 355 (28) | 416 (27)
Statistical Analysis 1: Comparison: Part 2: Morphine vs Part 2: Morphine and Single Dose Cannabidiol; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.13, Mixed Models Analysis; Analyses are not adjusted for multiplicity; Geometric mean ratio = 1.08, 90% CI 2-sided [0.99 to 1.18] — Comparison was the effect of a single dose of cannabidiol on morphine compared to morphine alone
Statistical Analysis 2: Comparison: Part 2: Morphine vs Part 2: Morphine and Multiple Doses of Cannabidiol; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < 0.01, Mixed Models Analysis; Analyses are not adjusted for multiplicity; Geometric mean ratio = 1.26, 90% CI 2-sided [1.17 to 1.36] — Comparison was the effect of multiple doses of cannabidiol on morphine compared to morphine alone

15. Secondary Outcome: Part 2 - M6G Cmax When Morphine is Administered Alone Versus When Co-administered With Cannabidiol.
Description: Cmax will be determined by collecting pharmacokinetic (PK) blood samples and calculated using noncompartmental analysis.13 PK samples will be obtained with each morphine dose for a total number of 39 PK samples per morphine cohort participant. The outcome measure reported will be the geometric mean ratio for morphine-6-glucuronide (M6G) alone compared to morphine-6-glucuronide (M6G) after 7 days of CBD dosing.
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 12, 24, and 48 hours after each morphine dose (Days 1, 4, and 11)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2: Morphine | Part 2: Morphine and Single Dose Cannabidiol | Part 2: Morphine and Multiple Doses of Cannabidiol
Number analyzed (Participants) | 20 | 20 | 18
ng/mL | 47 (24) | 51 (28) | 52 (28)
Statistical Analysis 1: Comparison: Part 2: Morphine vs Part 2: Morphine and Single Dose Cannabidiol; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.12, Mixed Models Analysis; Analyses are not adjusted for multiplicity; Geometric mean ratio = 1.08, 90% CI 2-sided [1.00 to 1.17] — Comparison was the effect of a single dose of cannabidiol on morphine compared to morphine alone
Statistical Analysis 2: Comparison: Part 2: Morphine vs Part 2: Morphine and Multiple Doses of Cannabidiol; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.07, Mixed Models Analysis; Analyses are not adjusted for multiplicity; Geometric mean ratio = 1.11, 90% CI 2-sided [1.01 to 1.21] — Comparison was the effect of multiple doses of cannabidiol on morphine compared to morphine alone

ADVERSE EVENTS:
Time Frame: Part 1: 36 days Part 2: 24 days
Arm/Group | Cannabidiol (Part 1) | Placebo (Part 1) | Cannabidiol and Citalopram Drug Interaction (Part 2) | Cannabidiol and Morphine Drug Interaction (Part 2)
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/50 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/50 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 43/151 | 9/50 | 7/20 | 5/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cannabidiol (Part 1) (N=151) | Placebo (Part 1) (N=50) | Cannabidiol and Citalopram Drug Interaction (Part 2) (N=20) | Cannabidiol and Morphine Drug Interaction (Part 2) (N=20)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Application Site Irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod Bite (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacterial Vaginosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 0 (0) | 2 (3) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Dry Mouth (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Epigastric Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 4 (4) | 0 (0) | 2 (3) | 0 (0)
Hepatic Enzyme Increase (Hepatobiliary disorders) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Lymphadenopathy Cervical (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nightmares (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (General disorders) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
Urine Odor Foul (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urogenital Trichomoniasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venipuncture Site Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral Syndrome (Infections and infestations) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Distention (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling Hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Abrasion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal Burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 serology test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Decreased Appetite (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Non-sustained ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/89/NCT06192589/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT06192589/SAP_001.pdf
  • Informed Consent Form (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT06192589/ICF_002.pdf